CLINICAL TRIAL: NCT02498691
Title: Perinatal Consequences of Endometriosis: Multicenter Prospective Comparative Study
Brief Title: Perinatal Consequences of Endometriosis
Acronym: ENDOBST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P140304
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis
Keywords: endometriosis; preterm delivery; caesarean; Pregnancy outcomes of women with or without endometriosis
MeSH Terms: conditions — Endometriosis; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type exposed (Experimental): endometriosis
  Interventions: Biological: Biological collection
- Type unexposed (Experimental): Without endometriosis
  Interventions: Biological: Biological collection

INTERVENTIONS:
Biological: Biological collection — Blood and saliva samples, placenta and cord blood collection

SUMMARY:
Endometriosis is a benign gynecological disease, characterized by the presence of endometrium-like tissue outside the uterine cavity that affect up to 10-15% of women in reproductive age worldwide, with an extensive impact on women's wellbeing and their reproductive life. Endometriosis lesions are heterogeneous and three phenotypes of the disease are well recognized and are fundamentally different from each other: superficial peritoneal endometriosis (peritoneal implants), ovarian endometrioma (cyst ovarian endometriosis), and deeply infiltrating endometriosis (invasive nodules greater than 5 mm).

The investigators performed a prospective multicenter comparative study to assess the maternal and fetal risks related to endometriosis during pregnancy, regarding disease phenotype, This study will evaluate with sufficient power the risk of prematurity and obstetrical complications associated with endometriosis according to disease phenotype.

This study aims to provide new informations to pregnant women with endometriosis, guide the monitoring of pregnancy, optimize management strategies based on the nature of complications and ultimately to improve the health of women and their unborn child

DETAILED DESCRIPTION:
Design selected and justification: the study ENDOBST is a

* exposed / unexposed type
* in superiority
* with two comparative groups (endometriosis / without endometriosis)
* Ratio of distribution of subjects in study groups = 1: 2

ENDOBST is a comparative prospective multicenter study presentation exposed - unexposed type. The study aims to compare the outcomes of pregnancy in the whole exposed group to controls and then according to the three disease phenotype (superficial, ovarian, and deep endometriosis).

Endobst aims to test the hypothesis that women with endometriosis have an increased risk of preterm delivery (primary endpoint) and an increased risk of pregnancy complications (secondary endpoints) when compared to diseases-free women. Comparisons will be performed according to disease phenotype.

These analyzes will be conducted after taking into account factors likely to influence the occurrence of preterm birth such as particularly social characteristics (education level, employment status), age and body mass index of women, pathological medical and obstetrical history and behavioral factors (tobacco).

Secondary analyzes will be conducted to investigate the link between endometriosis, and other adverse pregnancy outcomes (premature rupture of membranes, intrauterine growth restriction), complications related to the surgical treatment endometriosis prior to pregnancy.

Regarding the previous surgical treatment, the subgroup of women operated for their endometriosis will be compared to the subgroup of non-operated endometriosis in women and free subset of women. Particular attention will be paid to the phenotype of endometriosis and the nature of previous surgical treatment for pregnancy to control bias indication inherent in observational studies. These associations will be studied from multivariate regression models.

ELIGIBILITY:
Inclusion Criteria:

* Patient major
* Single Pregnancy
* Patient followed before 22 SA and giving birth in the maternity ward in the study
* Affiliated to health care

Exclusion Criteria:

* Opposition to the use of personal medical data or medical data of their child for research purposes
* Pregnant women with multiple pregnancies
* HIV positive women
* Patients addressed in the center as part of a transfer in utero.
* Women whose pregnancy is complicated by a spontaneous miscarriage before 15 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1444 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Number of preterm delivery | at Day 0 until 26 weeks
  Each delivery greater than or equal to 22 weeks and less than 37 weeks

SECONDARY OUTCOMES:
premature rupture of membranes | at Day 0 until 26 weeks
fetal loss | at Day 0 until 11 weeks
intrauterine growth restriction | at Day 0 until 31 weeks
induced or spontaneous preterm birth | at Day 0 until 26 weeks
preeclampsia | at Day 0 until 31 weeks
placenta previa | at Day 0 until 31 weeks
postpartum hemorrhage | at 11 weeks until 31 weeks
number of caesarean | at 11 weeks until 31 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Chapron, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Francois Goffinet, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcellin L, Goffinet F, Azria E, Thomin A, Garabedian C, Sibiude J, Verspyck E, Koskas M, Santulli P, Rousseau J, Ancel PY, Chapron C. Association Between Endometriosis Phenotype and Preterm Birth in France. JAMA Netw Open. 2022 Feb 1;5(2):e2147788. doi: 10.1001/jamanetworkopen.2021.47788. PMID 35133433